CLINICAL TRIAL: NCT03494114
Title: Imaging Activated Macrophages in the Lungs
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding has ended and unable to recruit due to COVID 19
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Endocyte (Industry)
Responsible Party: Principal Investigator, Timothy Blackwell, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 180071
Record Dates: First submitted 2018-03-15; First posted 2018-04-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Testing whether folate-based imaging using 68 Ga-EC2115 can be used to identify macrophages expressing the high affinity folate receptor (folate receptor beta).
Who Masked: Outcomes Assessor
Masking Description: The radiologist who evaluates the PET scan will be blinded to the to patient groups (COPD versus control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COPD Patients (Experimental): Folate imaging will be performed with 68Ga-EC2115 prior to scheduled bronchoscopy, which will be performed for clinical purposes to evaluate a suspicious lung nodule. The unused portion of the bronchoalveolar lavage (not necessary for clinical purposes), will be interrogated to compare PET imaging with parameters of inflammation in BAL, including the number/percentage of macrophages expressing FRβ. In addition, PET imaging data will be compared with disease severity, based on pulmonary function testing.
  Interventions: Drug: Ga-EC2115
- Individuals without COPD (Experimental): Folate imaging will be performed with 68Ga-EC2115 prior to scheduled bronchoscopy, which will be performed for clinical purposes to evaluate a suspicious lung nodule. The unused portion of the bronchoalveolar lavage (not necessary for clinical purposes), will be interrogated to compare PET imaging with parameters of inflammation in BAL, including the number/percentage of macrophages expressing FRβ.
  Interventions: Drug: Ga-EC2115

INTERVENTIONS:
Drug: Ga-EC2115 — Ga-EC2115 will be administered by IV injection prior to PET/CT imaging.

SUMMARY:
To test whether folate-based positron emission tomography (PET) imaging using 68Ga-EC2115 can differentiate chronic obstructive pulmonary disease (COPD) patients from control subjects and determine whether the PET signal correlates with measurements of inflammation and disease severity.

DETAILED DESCRIPTION:
Investigators intend to enroll patients who are undergoing bronchoscopy for diagnosis of solitary pulmonary nodules from the Vanderbilt lung nodule evaluation clinic, including 30 patients with COPD and 15 patients without COPD. Folate imaging will be performed with 68Ga-EC2115 within one week prior to scheduled bronchoscopy or from 1 week to 6 months after scheduled bronchoscopy, which will be performed for clinical purposes. The unused portion of the bronchoalveolar lavage (not necessary for clinical purposes), will be interrogated to compare PET imaging with parameters of inflammation in bronchoalveolar lavage (BAL). In addition, PET imaging data will be compared with disease severity based on pulmonary function testing.

ELIGIBILITY:
Inclusion Criteria:

* ≥45 years of age
* Pulmonary function testing done within last 2 years

  * For COPD group, forced expiratory volume at one second/forced vital capacity (FEV1/FVC) ratio < 0.7 and FEV1 < 80% predicted.
  * For control group, FEV1/FVC ratio > 0.7 and FEV1 > 80% predicted.
* Scheduled to undergo bronchoscopy for diagnostic evaluation of solitary pulmonary nodule (< 3 cm in diameter)

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant or lactating women. (Serum pregnancy testing will be required for pre-menopausal women within 24 hours of PET scanning)
* Diagnosis of chronic lung disease other than COPD, i.e. - asthma, idiopathic pulmonary fibrosis
* History of diagnosis or treatment of lung cancer

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Determine whether the PET signal in the lungs correlates with inflammation in bronchoalveolar lavage (BAL). | 1 day (at the time of bronchoscopy following PET scanning)
  We will compare the PET signal from 68 Ga-EC2115 in the lungs (opposite lung to the one containing a lung nodule) to the number of macrophages and other inflammatory cells obtained by BAL, particularly those expressing folate receptor beta.

SECONDARY OUTCOMES:
Determine whether the PET signal in lungs can identify differences between patients with COPD and control subjects without COPD. | 1 day (at the time of the PET scan)
  We will compare the PET signal from 68 Ga-EC2115 in the lungs (opposite lung to the one containing a lung nodule) of patients with COPD and control subjects without COPD (based on pulmonary function testing).

OTHER OUTCOMES:
Determine whether the PET signal in lungs correlates with COPD severity. | 1 day (at the time of the PET scan)
  We will compare the PET signal from 68 Ga-EC2115 in the lungs (opposite lung to the one containing a lung nodule) of COPD patients and determine whether there is a correlation between PET signal and severity of COPD based on FEV1 (percent of predicted).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Blackwell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No